CLINICAL TRIAL: NCT00956540
Title: Effect of Deflating the Tracheal Cuff During Ventilatory Disconnections on Weaning Time
Brief Title: Does Deflating the Tracheal Cuff Shorten Weaning Time?
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital Virgen de la Salud (Other)
Responsible Party: Principal Investigator, Gonzalo Hernandez Martinez, FEA Medicina Intensiva, Hospital Virgen de la Salud
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 29/06/09-54
Record Dates: First submitted 2009-08-06; First posted 2009-08-11 (Estimated); Results first posted 2011-09-27 (Estimated); Last update posted 2011-09-27 (Estimated); Status verified 2011-08

CONDITIONS: Weaning; Tracheostomy
Keywords: Tracheostomy; decannulation; weaning; Tracheostomy Weaning

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Deflating (Experimental): Deflating tracheal cuff (total air suction under negative pressure using a syringe) during periods of disconnection from mechanical ventilation in the weaning phase in patients tracheostomized for prolonged weaning or ventilatory support. During ventilatory support the tracheal cuff remain pressurized (30 mmHg).
  Interventions: Procedure: Deflating tracheal cuff
- Not deflating (No Intervention): The tracheal cuff remain inflated all the time during the weaning phase in patients tracheostomized for prolonged weaning or ventilatory support
- Deflating 2 (Experimental): Deflating tracheal cuff during periods of disconnection from mechanical ventilation in the weaning phase in patients tracheostomized for low level of consciousness or inability to adequate mange the airway.
  Interventions: Procedure: Deflating tracheal cuff 2
- Not deflating 2 (No Intervention): The tracheal cuff remain inflated all the time during the weaning phase in patients tracheostomized for low level of consciousness or inability to adequate mange the airway.

INTERVENTIONS:
Procedure: Deflating tracheal cuff — Deflating tracheal cuff during ventilatory disconnections along the weaning phase in patients tracheostomized for prolonged weaning or ventilatory support.
  Arms: Deflating
Procedure: Deflating tracheal cuff 2 — Deflating tracheal cuff during ventilatory disconnections along the weaning phase in patients tracheostomized for low level of consciousness or inability to adequate manage the airway.
  Arms: Deflating 2

SUMMARY:
The purpose of this study is to determine whether deflating the tracheal cuff in tracheostomized patients, during disconnections from ventilatory support along the weaning phase shortens the weaning time.

DETAILED DESCRIPTION:
Randomized controlled trial.

Study protocol: patients will be eligible for the study after fulfilling standard criteria for weaning initiation and stratified for risk of aspiration (drink test)into two categories:

* Low/moderate risk patients (see later).
* High risk patients (spontaneous aspiration of pharyngeal secretions), will be excluded from the study.

After this evaluation patients will be randomized (concealed allocation) stratifying with the tracheostomy indication.

Weaning and Decannulation Protocol: Attempts to discontinue mechanical ventilation (MV) will be initiated when the tracheostomized patients fulfill the criteria (recovery from the precipitating illness; respiratory criteria consisting of a PaO2/fraction of inspired oxygen ratio of >150 mm Hg with a positive end-expiratory pressure <8 cm H2O, and an arterial pH >7.32; and clinical criteria consisting of the absence of myocardial ischemia determined by ECG, no need for vasoactive drugs or dopamine ≤5 µg/kg/min, a heart rate <140 beats/min, haemoglobin concentration >8 g/dL, temperature <38°C, no need for sedative drugs, presence of respiratory stimulus and spontaneous cough deemed clinically appropriate. Patients will be screened daily for these criteria).

A clinical algorithm for progressive weaning from mechanical ventilation will be followed at the discretion of the attending physician. Patients will be weaned following one of two methods: progressive withdrawal of pressure support ventilation or T-tube trials. When patients tolerate spontaneous breathing for 12 hours on two consecutive days, they will remain connected to the T-tube continuously.

When the patient remain disconnected from mechanical ventilation for at least 24 hours, the investigators will assess his or her preparedness for decannulation. The investigators will perform the tracheostomy tube occlusion test to exclude tracheal obstruction to airflow.

At this point, the attending physician clinically will evaluate the patient's capacity to clear respiratory secretions mainly based on the frequency of the need for suctioning and the characteristics of respiratory secretions.

The nurse will suction subglottic secretions while deflating the cuff to avoid the risk of aspiration.

Criteria for decannulation: respiratory secretions management considered adequate (<2 aspiration every 8 hours) and low risk of aspiration.

End-points:

* Weaning time: starting the day of first disconnection (lasting <30 minutes)and ending the day the patient is liberated from mechanical ventilation (patients will be considered weaned after 24 consecutive hours disconnected from mechanical ventilation).
* Tracheobronchitis and pneumonia after randomization. Safety considerations: The main safety concern is the risk of aspiration. First all patients will be categorized in three steps using the drink test: low risk patients (normal drink test) with no other specific interventions; moderate risk (abnormal drink test) the risk of aspiration study will include a videolaryngoscopy; high risk patients will be excluded from the study. In all patients a high flow-humidified oxygen-air mixture system will be connected trough the external cannula.

ELIGIBILITY:
Inclusion criteria: tracheostomized patients for any of the following reasons:

* Prolonged time under mechanical ventilation (>21 days) or prolonged weaning.
* Motor component of Glasgow Coma Score <6 points or inability to adequate manage the airway (>2 aspirations every 8 hours).

Exclusion Criteria:

* High risk of aspiration (neuromuscular disease affecting bulbar functions, tracheostomies indicated as a part of a surgical procedure involving the upper airway or high risk of aspiration observed after specific evaluation previous to randomization).
* Death before starting weaning attempts.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 195 (Actual)
Dates: Start 2009-12; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gonzalo Hernandez, MD, Study Chair — Hospital Virgen de la Salud; Maria del Mar Cruz, MD, Principal Investigator — Hospital Virgen de la Salud
Locations (1):
- Hospital Virgen de la Salud, Toledo, Toledo, Spain

REFERENCES:
- [Derived] Hernandez G, Pedrosa A, Ortiz R, Cruz Accuaroni Mdel M, Cuena R, Vaquero Collado C, Garcia Plaza S, Gonzalez Arenas P, Fernandez R. The effects of increasing effective airway diameter on weaning from mechanical ventilation in tracheostomized patients: a randomized controlled trial. Intensive Care Med. 2013 Jun;39(6):1063-70. doi: 10.1007/s00134-013-2870-7. Epub 2013 Mar 8. PMID 23471512

RESULTS

PARTICIPANT FLOW:
Groups:
- Deflating: The tracheal cuff is deflating during disconnection from mechanical ventilation periods in patients tracheostomized for prolonged weaning or ventilatory support. While patients are connected to mechanical ventilation, the cuff is reinflated.
- Not Deflating: The tracheal cuff remains inflated during disconnections from mechanical ventilation periods until the patients is definitively liberated from mechanical ventilation in patients tracheostomized for prolonged weaning or ventilatory support
- Deflating 2: The tracheal cuff is deflated during disconnections from mechanical ventilation periods in patients tracheostomized for low level of consciousness or inability to adequate mange the airway. The cuff is reinflated when the patients is connected to mechanical ventilation.
- Not Deflating 2: The tracheal cuff remains inflated during the weaning period until the patient is definitively liberated from mechanical ventilation in patients tracheostomized for low level of consciousness or inability to adequate manage the airway.
Period: Overall Study
Arm/Group | Deflating | Not Deflating | Deflating 2 | Not Deflating 2
Started | 54 | 50 | 46 | 45
Completed | 51 | 46 | 43 | 41
Not Completed | 3 | 4 | 3 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Deflating | Not Deflating | Deflating 2 | Not Deflating 2 | Total
Number analyzed (Participants) | 54 | 50 | 46 | 45 | 195
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 40 | 35 | 44 | 40 | 159
  >=65 years | 14 | 15 | 2 | 5 | 36
Age Continuous [Mean (Standard Deviation); unit: years] | 56 (16) | 58 (19) | 56 (16) | 58 (19) | 57 (17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 17 | 16 | 19 | 75
  Male | 31 | 33 | 30 | 26 | 120
Region of Enrollment [Number; unit: participants]
  Spain | 54 | 50 | 46 | 45 | 195

OUTCOME MEASURES:

1. Secondary Outcome: Tracheobronchitis and Pneumonia
Time Frame: 6 months
Reporting Status: Not Posted

2. Primary Outcome: Weaning Time
Description: The weaning time starts at the first disconnection from mechanical ventilation lasting >30 minutes and ends after the patient tolerate 24 consecutive hours disconnected from mechanical ventilation.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: day
Arm/Group | Deflating | Not Deflating | Deflating 2 | Not Deflating 2
Number analyzed (Participants) | 55 | 50 | 46 | 44
day | 4.95 (5) | 10.15 (10) | 4.95 (5) | 10.15 (10)

ADVERSE EVENTS:
Arm/Group | Deflating | Not Deflating | Deflating 2 | Not Deflating 2
Serious Adverse Events (participants affected / at risk) | 10/54 | 16/50 | 9/46 | 15/45
Other Adverse Events (participants affected / at risk) | 0/54 | 0/50 | 0/46 | 0/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Deflating (N=54) | Not Deflating (N=50) | Deflating 2 (N=46) | Not Deflating 2 (N=45)
respiratory infection (Infections and infestations) | 10 (10) | 16 (16) | 9 (9) | 15 (15)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No